CLINICAL TRIAL: NCT02676752
Title: Assessing Skin/Soft Tissue Elasticity in Head and Neck Cancer Survivors
Brief Title: Skin/Soft Tissue Elasticity in Head and Neck Cancer Survivors With Lymphedema and Fibrosis
Status: Completed | Type: Observational
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kenneth Niermann, Principal Investigator, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 15135; NCI-2016-00069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC HN 15135 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2016-02-03; First posted 2016-02-08 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Lymphedema
Keywords: head and neck cancer; lymphedema and fibrosis
MeSH Terms: conditions — Lymphedema; Head and Neck Neoplasms; Fibrosis | interventions — Independent Medical Evaluation; Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Skin/soft tissue elasticity assessment: Participants will be evaluated for LEF status using the HN-LEF Grading Criteria and neck range of motion using the Cervical Range of Motion Device. Participants also complete study questionnaires, including VHNSS and LSIDS-H&N. Participants undergo ultrasound shear wave elastography over 20-25 minutes. Participants' cancer disease and treatment information will be gathered from their medical records.
  Interventions: Procedure: Medical Examination; Other: Questionnaire Administration; Procedure: Shear Wave Elastography

INTERVENTIONS:
Procedure: Medical Examination — Evaluation of secondary lymphedema and fibrosis (LEF) status
  Other Names: Exam; Examination; Medical Assessment; Medical Exam; Medical Inspection
Other: Questionnaire Administration — Completion of questionnaires
Procedure: Shear Wave Elastography — Undergo ultrasound shear wave elastrography
  Other Names: Transient Elastography

SUMMARY:
This research trial studies skin/soft tissue elasticity in head and neck cancer survivors with lymphedema and fibrosis. Lymphedema and fibrosis is a common effect of head and neck cancer which may lead to skin tightness, pain, and body image issues. Early detection of lymphedema and fibrosis may help reduce serious functional loss of the neck. Shear wave elastography is a technique that provides a quantitative measure of stiffness using a push pulse to generate shear waves within the tissues. Conventional imaging techniques are then used to monitor the shear waves generated through the tissue to calculate the shear wave speed. Shear wave elastography may help obtain an early and accurate measurement of tissue elasticity in head and neck cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain pilot data of the elasticity of skin/soft tissues using shear wave elasticity at the defined anatomical sites in head and neck cancer survivors with lymphedema and fibrosis (LEF).

II. To explore the correlation between elasticity of skin/soft tissues and the following: 1) symptoms as measured by the Lymphedema Symptom Intensity and Distress Survey-Head and Neck (LSIDS-HN); 2) functional impact as measured by Cervical Range of Motion Device and the Vanderbilt Head and Neck Symptom Survey; and 3) physical exam findings as measured by Head and Neck LEF Grading Criteria.

OUTLINE:

Participants will be evaluated for LEF status using the Head and Neck External Lymphedema - Fibrosis (HN-LEF) Grading Criteria and neck range of motion using the Cervical Range of Motion Device. Participants also complete study questionnaires, including Vanderbilt Head and Neck Symptom Survey (VHNSS) and Lymphedema Symptom Intensity and Distress Survey - Head and Neck (LSIDS-H&N). Participants undergo ultrasound shear wave elastography over 20-25 minutes. Participants' cancer disease and treatment information will be gathered from their medical records.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed cancer involving the head and neck
* Completed all therapy
* No evidence of cancer (NED)
* Ability to understand English in order to complete questionnaires
* Able to provide informed consent

Exclusion Criteria:

* Have medical record documentation of significant cognitive impairment that would preclude the ability to provide informed consent
* Are unwilling to undergo the study assessment
* Have recurrent and/or metastatic cancer

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults 22 years and older that are head and neck cancer survivors and have lymphedema and fibrosis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Elasticity values | Within 2 weeks of initial study visit
  Descriptive statistics will be used to describe data from elasticity measure. Of particular interest will be the measures of central tendency and variability at the multiple sites. Sites with higher variability (coefficient of variation) that others may be indicative of less reliable assessment.

SECONDARY OUTCOMES:
Strength of associations of tissue elasticity and current conventional methods | Within 2 weeks of initial study visit
  Correlation coefficients will be used to assess the strength of the associations of the elasticity values with the respective LEF grades (HN-LEF) for the respective sites. Those values will also be correlated with Vanderbilt Head and Neck Symptom Survey and HN-LSIDS symptom and Cervical Range of Motion scores. Due to the large number of correlations proposed in this study, effect sizes (strength of the associations) and clinically significant patterns will be of much greater importance than statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Niermann, Principal Investigator — Vanderbilt University/Ingram Cancer Center
Locations (1):
- Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee, United States

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://vicc.org/ct/